CLINICAL TRIAL: NCT00678041
Title: A Randomized, Double-blind, Placebo-controlled Trial Examining the Effect of Nitrofurantoin Prophylaxis in Women Performing Clean Intermittent Self-catheterization (CISC) After Surgery for Urinary Incontinence and/or Pelvic Organ Prolapse
Brief Title: Nitrofurantoin and Urinary Tract Infections (UTIs)
Acronym: APPIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient recruitment
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Gary Sutkin, Physician, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SutkinAppic
Record Dates: First submitted 2008-05-10; First posted 2008-05-15 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Tract Infections
Keywords: urinary catheterization; urinary tract infection; urinary incontinence; pelvic floor prolapse; antibiotics
MeSH Terms: conditions — Urinary Tract Infections; Urinary Incontinence | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Nitrofurantoin Group (Experimental): extended release nitrofurantoin 100mg to be taken daily while performing clean intermittent self-catheterization (CISC) and for three more days after stopping CISC
  Interventions: Drug: Nitrofurantoin
- Arm 2: Placebo Group (Placebo Comparator): identical appearing placebo capsule to be taken daily while performing clean intermittent self-catheterization (CISC) and for three more days after stopping CISC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrofurantoin — nitrofurantoin 100mg to be taken daily while performing clean intermittent self-catheterization (CISC) and for three more days after stopping CISC
  Other Names: Macrodantin
  Arms: Arm 1: Nitrofurantoin Group
Drug: Placebo — Placebo capsule to be taken daily while performing clean intermittent self-catheterization (CISC) and for three more days after stopping CISC
  Arms: Arm 2: Placebo Group

SUMMARY:
Urinary tract infection (UTI) is the most common complication after surgery for prolapse or urinary incontinence. UTIs are painful and have the potential to turn into kidney infections. We are asking women who self-catheterize after surgery to try either an antibiotic or a placebo pill so we can see if we can prevent UTIs without causing side effects.

This study will not require any additional visits or blood draws. You will be asked to answer some questions, keep a brief diary of your experience, and immediately report any symptoms of a UTI to your doctor.

DETAILED DESCRIPTION:
Abstract:

Specific aim: to determine if extended release nitrofurantoin antibiotic prophylaxis administered to patients performing clean intermittent self-catheterization (CISC) after pelvic organ prolapse and/or urinary incontinence surgery decreases the incidence of symptomatic urinary tract infection (UTI) compared with placebo.

Study Design: Randomized double-blind placebo-controlled trial.

Methods: Consented patients who undergo urogenital surgery and fail their post-operative voiding trial will be randomized to either extended release nitrofurantoin 100mg or an identical appearing placebo capsule to be taken daily while performing CISC and for three subsequent days after stopping CISC. Catheterized urine specimens will be sent for culture and sensitivity when women report symptoms consistent with cystitis. Symptomatic UTI will be defined using strict culture-based definitions. We anticipate that the study will end within 6 weeks of starting CISC.

Data Analysis: Primary and secondary outcomes will be evaluated with Student t test and Fisher exact test.

Sample Size: Assuming a decrease in symptomatic UTIs attributable to nitrofurantoin prophylaxis from 33% to 10%, with 80% power, and a two-sided alpha of 0.05, and a 10% dropout rate, we should recruit a total of 108 patients.

ELIGIBILITY:
Inclusion Criteria:

* Women who fail a post-operative voiding trial and are willing to learn clean intermittent self-catheterization (CISC) prior to discharge from the hospital

Exclusion Criteria:

* Known drug allergy to nitrofurantoin
* A history of renal insufficiency
* Renal transplant
* Renal nephropathy
* A recent history of more than 3 Urinary Tract Infections (UTIs) per year
* Known immunocompromised condition (organ transplant, chemotherapy for cancer or arthritis, autoimmune diseases (lupus etc)).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sutkin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a double blind 1:1 randomized trial
Groups:
- Arm 1: Nitrofurantoin Group: extended release nitrofurantoin 100mg to be taken daily while performing CISC and for three more days after stopping CISC
  Nitrofurantoin: nitrofurantoin 100mg to be taken daily while performing CISC and for three more days after stopping CISC
- Arm 2: Placebo Group: identical appearing placebo capsule to be taken daily while performing CISC and for three more days after stopping CISC
  Placebo: Placebo capsule to be taken daily while performing CISC and for three more days after stopping CISC
Period: Overall Study
Arm/Group | Arm 1: Nitrofurantoin Group | Arm 2: Placebo Group
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — Physician Decision | 5 | 5

BASELINE CHARACTERISTICS:
Population: This is a randomized, double-blind, placebo-controlled clinical trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nitrofurantoin Group | Arm 2: Placebo Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Customized [Number; unit: participants]
  at least 18 yrs of age | 5 | 5 | 10
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Symptomatic UTI's Confirmed With a Positive Urine Culture Within 6 to 8 Weeks After CISC Teaching and Implementation
Description: Participants are to be assessed for UTI systems and f/u urine culture routine over a period of 6 to 8 weeks after CISC teaching and implementation.
Time Frame: 6 to 8 weeks after surgery
Population: 0 participants analyzed due to study termination. Study terminated prior to accumulation of any data. Participating subjects were withdrawn prior to measuring any outcome data.
Arm/Group | Arm 1: Nitrofurantoin Group | Arm 2: Placebo Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time (Days After Surgery) to Development of Symptomatic, Culture Documented UTI
Description: 0 participants analyzed due to study termination. Study terminated prior to accumulation of any data. Participating subjects were withdrawn prior to measuring any outcome data.
Time Frame: 6 weeks after surgery
Population: as for outcome 1
Groups:
- All Patients: 0 participants analyzed due to study termination. Study terminated prior to accumulation of any data. Participating subjects were withdrawn prior to measuring any outcome data.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency of Urine Cultures Positive for Organism Strains That Are Resistant to Nitrofurantoin and Other Commonly Used Antibiotics.
Description: 0 participants analyzed due to study termination.Study terminated prior to accumulation of any data. Participating subjects were withdrawn prior to measuring any outcome data.
Time Frame: 6 weeks after surgery
Population: as for outcome 1
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Adherence to CISC
Description: as for outcome 2
Time Frame: 6 weeks after surgery
Population: as for outcome 1
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Patient Perceptions Regarding CISC
Description: as for outcome 2
Time Frame: 6 weeks after surgery
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Frequency of Adverse Events Related to CISC Such as Urethral Pain, Irritative Voiding Symptoms, Hematuria
Description: as for outcome 2
Time Frame: 6 weeks after surgery
Population: as for outcome 1
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Frequency of Adverse Events Related to Daily Nitrofurantoin Exposure Such as Nausea, Diarrhea, C. Difficile Colitis
Description: as for outcome 2
Time Frame: 6 weeks after surgery
Population: as for outcome 1
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data was collected from the point of surgery up to a period of 6 to 8 weeks post surgery and completion of CISC (Clean Intermittent Self-catheterization)
Arm/Group | Arm 1: Nitrofurantoin Group | Arm 2: Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Study terminated prior to accumulation of any data. Participating subjects were withdrawn prior to measuring any outcome data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes